CLINICAL TRIAL: NCT06066398
Title: Evaluation of Thoracoscopic Pleural Lavage and Pleural Brushing as Unconventional Methods for Diagnosis of Pleural Effusion
Brief Title: Thoracoscopic Pleural Lavage and Brushing in Undiagnosed Pleural Effusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Emad El-din Abdalah, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Thoraco pleural lavage & brush
Record Dates: First submitted 2023-09-06; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Disorder of Pleura and Pleural Cavity
MeSH Terms: conditions — Pleural Diseases

STUDY DESIGN:
Intervention Model Description: single group will be undergone thoracoscopy where pleural forceps biopsy, pleural brush and pleural lavage will be taken
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- medical thoracoscope (Other): medical thoracoscope will be done during which pleural brush, pleural forceps biopsy and pleural lavage will be taken to compare yield of diagnosis and safety between them
  Interventions: Procedure: medical thoracoscope; Diagnostic Test: Forceps biopsy and pleural brush histopathology; Diagnostic Test: pleural lavage cytology

INTERVENTIONS:
Procedure: medical thoracoscope — Medical thoracoscopy will be performed during which pleural brush will be used first followed by forceps biopsy to obtain pleural specimens from suspect areas under visual control and pleural lavage will be performed by injecting 300 mL of normal saline
Diagnostic Test: Forceps biopsy and pleural brush histopathology — Forceps biopsy and pleural brush will be obtained for histopathological examination for diagnosis
Diagnostic Test: pleural lavage cytology — pleural lavage will be obtained for cytological examination for diagnosis

SUMMARY:
1. To evaluate the diagnostic yield and safety of thoracoscopic pleural lavage and pleural brushing in cases of undiagnosed exudative pleural effusion.

DETAILED DESCRIPTION:
The diagnosis of etiology of pleural effusions remains a challenging issue even after diagnostic thoracocentesis and closed pleural biopsy in significant number of cases. In order to get a pleural biopsy or the diagnosis of undiagnosed pleural effusion, several techniques were used, such as percutaneous needle pleural biopsy, CT guided pleural biopsy, medical thoracoscopy, video-assisted thoracoscopy and open thoracotomy.

Medical thoracoscopy plays a huge role with a great diagnostic yield in the diagnosis of exudative pleural effusion. Pleural biopsy is considered to be a gold standard investigation of choice in patients with undiagnosed exudative pleural effusions. It can be used to describe the diagnostic and therapeutic exploration of the pleural space mostly under local anesthesia with or without conscious sedation, unlike video-assisted thoracoscopic surgery (VATS), which is conducted under general anesthesia with single lung ventilation.

Pleural biopsy with forceps is the usual mode of obtaining thoracoscopic specimens from suspected pleural lesions. However, this may be associated with complications like bleeding that hinders further biopsy, additionally, the decision to take biopsy could be difficult, especially when the targeted lesions are on the visceral pleura or near the vessels.

On the other hand, pleural brush could be used to safely obtain pleural specimens through medical thoracoscopy from suspected areas either in the parietal, visceral pleura or near the vascular structure.

The use of pleural lavage performed by injecting normal saline to pleural space and aspirated at the time of thoracoscopy would provide a higher diagnostic yield than the cytologic analysis of the fluid obtained at thoracentesis and could provide additional diagnostic information to thoracoscopic biopsy. This finding could be explained by one of the following:

1. The cells in the lavage are fresher and have not undergone degeneration as have many cells in the pleural fluid.
2. The lavage procedure could dislodge cells that would not have been detached otherwise. Tumor cells seeded in the subserous layer are exfoliated into the pleural cavity, and lavage could lead to the recovery of malignant cells.
3. Biopsies of the parietal and visceral pleura could have exposed the tumor and allowed malignant cells to be shed into the lavage fluid.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have documented exudative pleural effusion in whom the initial pleural tapping and closed pleural biopsy (CPB) will not be conclusive
* strong clinical and radiological data suggestive for alternative pathological diagnosis
* who will be admitted to our department

Exclusion Criteria:

* Patients with excess rib crowding with narrow inter-costal space and loculated pleural effusion cannot undergo thoracoscopy
* Patients with bleeding diathesis
* hemodynamic instability
* Arrhythmias
* intractable cough cannot be eligible to do thoracoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of efficacy which determined by the diagnostic yield | Baseline
  comparing thoracoscopic forceps biopsy, pleural brush and pleural lavage as regard efficacy which determined by the diagnostic yield

SECONDARY OUTCOMES:
Evaluation of safety which determined by occurance of complications | Baseline
  comparing thoracoscopic forceps biopsy, pleural brush and pleural lavage as regard safety which determined by occurance of complications

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sivagnaname Y-, Radhakrishnan P, Maria Selvam A. Thoracoscopic pleural brushing - an innovative method of pleural sampling in diagnostic medical thoracoscopy. Adv Respir Med. 2019;87(5):257-260. doi: 10.5603/ARM.2019.0046. PMID 31680224
- [Background] Bejui-Thivolet F, Guerin JC, Salle M, Milox A, Champel F, Vitrey D. [Thoracoscopy with pleural brushing. A new diagnostic method for pleural diseases]. Rev Pneumol Clin. 1984;40(5):311-9. French. PMID 6522932
- [Background] Bejui-Thivolet F, Guerin JC, Salle M, Milox A, Champel F, Vitrey D. [Contribution of thoracoscopic brushing to the diagnosis of pleural diseases]. Ann Pathol. 1984 Jun-Aug;4(3):195-201. French. PMID 6089845
- [Background] Blanc FX, Atassi K, Bignon J, Housset B. Diagnostic value of medical thoracoscopy in pleural disease: a 6-year retrospective study. Chest. 2002 May;121(5):1677-83. doi: 10.1378/chest.121.5.1677. PMID 12006460
- [Background] Mohamed KH, Mobasher AA, Yousef AI, Salah A, Ramadan MA, Emam AK, Alhayawan HM, Light RW. Pleural lavage: a novel diagnostic approach for diagnosing exudative pleural effusion. Lung. 2000 Nov-Dec;178(6):371-9. doi: 10.1007/s004080000040. PMID 11361060